CLINICAL TRIAL: NCT03492515
Title: A Multicenter Clinical Study of Recombinant Human Thrombopoietin(rhTPO) in Pregnancy With Immune Thrombocytopenia
Brief Title: Recombinant Human Thrombopoietin(rhTPO) in Pregnancy With Immune Thrombocytopenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: Peking University People's Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Linyi People's Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Shandong Provincial Hospital (Other Government); Zhongshan Bo Ai Hospital (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rhTPO in pregnancy of ITP
Record Dates: First submitted 2018-03-26; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Immune Thrombocytopenia
Keywords: immune thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group (Experimental): Accepting the treatment of rhTPO according platelet and bleeding condition
  Interventions: Drug: recombinant human thrombopoietin
- non-administered group (Active Comparator): No rhTPO will be used. If necessary, the patients will be given transfusion of platelets according to the their conditions.
  Interventions: Drug: Platelet Concentrate
- healthy control group (No Intervention): Healthy pregnant women and no use of any medicine。

INTERVENTIONS:
Drug: recombinant human thrombopoietin — If platelet count <30×10^9/L and with haemorrhage or risk of bleeding,the patients began to receive subcutaneous injection of TPO with the dose of 300 Unit/kg qd,duration ≤14 days;If platelet count is between 30×10^9/L and 50×10^9/L, the dose will be 300 Unit/kg qod;If platlet count ≥100×109/L, stop this treatment;After delivery, if platelet count <30×10^9/L and with haemorrhage or risk of bleeding,subcutaneous injection of TPO with the dose of 300 Unit/kg qd or qod will be given at a duration ≤14 days;If platelet count is between 30×10^9/L and 50×10^9/L, the dose will be 300 Unit/kg qw;If platlet count ≥100×109/L, stop the treatment.
  Other Names: rhTPO
  Arms: experimental group
Drug: Platelet Concentrate — according to the their conditions, use if necessary
  Arms: non-administered group

SUMMARY:
The purpose of this study was to observe the clinical efficacy and adverse reactions of rhTPO in the treatment of pregnancy-induced thrombocytopenia.

DETAILED DESCRIPTION:
The project is undertaken by Qilu Hospital of Shandong University and other 6 well-known hospitals in China. The investigators anticipate to undertaking a concurrent control, multicentre trial including 60 pregnancy associated ITP adult patients which are ineffective for first-line treatment or platelets infusion and 30 healthy pregnancy control. 30 of the ITP patients are selected to receive rhTPO(given different dose according to the platelet count, the risk of bleeding and delivery), the other ITP patients are selected not to receive rhTPO. Platelet count, bleeding and other symptoms of ITP patients and their newborns are evaluated after treatment, adverse events are also recorded throughout the study in order to report the efficacy and safety of the rhTPO for the treatment of pregnancy with ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. 18-50 years of age; gestational age over 32 weeks;
3. No response to the treatment of glucocorticoids and / or intravenous immunoglobulin (a stable dose of glucocorticoid could be accepted);
4. Platelet transfusion was not effective.
5. Platlet count of the patients <30* 10^9/L and had the risk of bleeding or bleeding.
6. No obvious abnormalities in liver and kidney function had (1.5 times higher than normal limit of the serum urea nitrogen, creatinine, serum transaminase and bilirubin );
7. No severe cardiac and pulmonary dysfunction;
8. No history of mental illness;
9. Voluntarily signed written informed consent.

Exclusion Criteria:

1. A history of serious allergies to biologics;
2. The history of thrombosis;
3. Thromboembolic or hemorrhagic disease;
4. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Platelet count during delivery | up to 2 years per subject
  Platelet count during delivery will be assessed

SECONDARY OUTCOMES:
Adverse events in neonates | up to 2 years per subject
  The number and frequency of therapy associated adverse events in neonates
platlet count of newborns | up to 42 days per newborn
  Platelet counts of D1, 3, and 7 of newborns, extended to d42 if thrombocytopenia occurs.
Adverse events in parturients | up to 2 years per subject
  The number and frequency of therapy associated adverse events in parturients

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou,, Dr, Principal Investigator — Shandong University
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No